CLINICAL TRIAL: NCT06041490
Title: A Randomized, Controlled, Open-label, Multi-center Clinical Trial of Multi-kinase Inhibitor Combined With Bevacizumab as Adjuvant Therapy in Patients With Hepatocellular Carcinoma and High-risk Recurrence Factors After Liver Transplantation
Brief Title: Adjuvant Therapy for High-risk Hepatocellular Carcinoma Post Liver Transplantation
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K4001
Record Dates: First submitted 2023-08-30; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-08

CONDITIONS: Liver Transplant; Complications; Hepatocarcinoma; Recurrent Osteosarcoma; High-Risk Cancer
Keywords: Hepatocarcinoma; Liver Transplant; Recurrence; High-Risk; multikinase inhibitor; bevacizumab
MeSH Terms: conditions — Carcinoma, Hepatocellular; Osteosarcoma; Recurrence | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- multi-kinase inhibitors in combination with bevacizumab (Experimental): TKI (Sorafenib 400mg, bid, po or Lenvatinib 8mg, qd, po if bodyweight less than 60 kg,12mg, qd, po if bodyweight more than 60kg or Donafenib：200mg, bid, po) + bevacizumab：7.5mg/kg, infusion, Q3w
  Interventions: Drug: multi-kinase inhibitors in combination with bevacizumab
- Without adjuvant therapy (No Intervention): No intervention.

INTERVENTIONS:
Drug: multi-kinase inhibitors in combination with bevacizumab — The eligible participants will start taking multi-kinase inhibitors between 4-8 weeks after liver transplantation. The choice of the specific multi-kinase inhibitor, including sorafenib, lenvatinib, or regorafenib, will be determined by the researchers based on factors such as the participant's tumor characteristics, liver function, physical condition, risk of side effects, economic status, and personal preference. The specific dosage and administration details can be found in the table provided. The maximum duration of multi-kinase inhibitor treatment will be 12 months or until any of the following conditions occur, whichever comes first: 1) The participant experiences intolerable toxic reactions that do not alleviate with dose adjustments, or 2) The participant has documented disease recurrence confirmed through imaging or withdraws from the study for other reasons.
  Arms: multi-kinase inhibitors in combination with bevacizumab

SUMMARY:
1. Explore the impact of postoperative administration of multi-kinase inhibitors (including sorafenib, lenvatinib, and regorafenib) in conjunction with bevacizumab on post-transplant recurrence, overall survival, and drug safety in liver transplant recipients at high risk of recurrence in hepatocellular carcinoma.
2. The primary objective of this study is to evaluate the efficacy of multi-kinase inhibitors in combination with bevacizumab as adjuvant therapy in liver transplant recipients with hepatocellular carcinoma who present high-risk factors for recurrence, based on the one-year recurrence-free survival rate (1-year RFS rate).
3. The secondary objectives of this study are to assess the effectiveness and safety of multi-kinase inhibitors in combination with bevacizumab as adjuvant therapy in liver transplant recipients with hepatocellular carcinoma who present high-risk factors for recurrence, based on the following parameters: Recurrence-free survival (RFS) duration, Overall survival (OS), Two-year and three-year RFS rates, Graft survival, Quality of life evaluation (QoL), Incidence of adverse events and serious adverse events.

DETAILED DESCRIPTION:
To investigate the effect of multikinase inhibitors (including sorafenib, lenvatinib and donafinib) combined with bevacizumab on recurrence, survival and safety in patients with hepatocellular carcinoma (HCC) at high risk of recurrence after liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary enrollment, accompanied by the signing of a written informed consent form, is a prerequisite for participation in this study. This ensures that participants enter the study based on their own decision and understanding of the research objectives, procedures, and potential risks.
2. The study includes individuals aged between 18 and 75 years, inclusive, without any gender restrictions. This broad age range and gender inclusivity allow for a diverse representation of participants, facilitating a comprehensive understanding of the study outcomes across different demographic profiles.
3. Prior to enrollment, participants must have undergone liver transplantation within the preceding 4 to 8 weeks. This specific time frame serves as an inclusion criterion to ensure that participants have recently undergone the surgical procedure, enabling researchers to investigate the effects of the transplantation within a relevant timeframe.
4. Participants must have a confirmed pathological diagnosis of hepatocellular carcinoma (HCC) and meet at least one of the following criteria:

   a) Pre-operative imaging or post-operative pathological confirmation of exceeding the Milan criteria.

   b) Presence of major vascular invasion. c) Post-operative pathological confirmation of the presence of microvascular invasion (MVI).

   d) Pre-operative imaging or post-operative pathological confirmation of the presence of satellite nodules.

   e) Recurrence of HCC after liver resection and subsequent liver transplantation.
5. Participants should have an anticipated life expectancy of more than 3 months.
6. Participants should not have received systemic anti-tumor treatment prior to liver transplantation, with the exception of pre-operative transarterial chemoembolization (TACE), traditional Chinese medicine, and interferon treatment.
7. Participants should have an Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1, indicating good functional status.
8. Participants' liver function, as assessed by the Child-Pugh score, should be classified as Grade A, indicating well-preserved liver function.
9. HBsAg-positive patients should receive continuous antiviral therapy post-transplantation, using first-line antiviral drugs such as entecavir, tenofovir, or tenofovir alafenamide.
10. Participants should have adequate hematological and organ function, based on the laboratory test results obtained within 14 days before the initiation of the study treatment, as follows:

    Laboratory tests (unless otherwise specified, no blood transfusion or use of G-CSF within 14 days prior to screening):
    1. Hemoglobin ≥ 90 g/L.
    2. White blood cell count ≥ 3.0 x 10^9/L.
    3. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L.
    4. Platelet count ≥ 75 x 10^9/L.

       Biochemical tests (no use of albumin within 14 days prior to screening):
    5. Serum albumin ≥ 28 g/L.
    6. Total bilirubin ≤ 2 times the upper limit of normal (ULN).
    7. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5 times ULN.
    8. Alkaline phosphatase (ALP) ≤ 5 times ULN.
    9. Creatinine ≤ 1.5 times ULN or creatinine clearance (CrCl) > 50 mL/min (calculated using the standard Cockcroft-Gault formula):

       - For females: CrCl = ((140 - age) x body weight (kg) x 0.85) / (72 x serum creatinine [mg/dL]).
       * For males: CrCl = ((140 - age) x body weight (kg) x 1.00) / (72 x serum creatinine [mg/dL]).

       Coagulation Function:
    10. International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 times the Upper Limit of Normal (ULN) or PT prolongation ≤ 6 seconds.
    11. Activated Partial Thromboplastin Time (APTT) ≤ 1.5 times ULN.
11. Women of Childbearing Potential: Women who agree to abstain from heterosexual intercourse during the treatment period and for at least 6 months after the last dose of the study drug, or use a contraceptive method with a failure rate of less than 1% per year. For women who have experienced menstrual bleeding and have not reached a postmenopausal state (continuous absence of menstruation for ≥12 months without any other known cause) and have not undergone sterilization procedures (removal of ovaries and/or uterus), they are considered to be of childbearing potential.

    1. Examples of contraceptive methods with a failure rate of less than 1% per year include bilateral tubal ligation, male sterilization, hormone-based contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
    2. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial, patients' preferred lifestyle, and daily activities. Periodic abstinence methods (such as calendar-based methods, ovulation period methods, symptothermal methods, or post-ovulation methods) and withdrawal are not acceptable contraceptive methods.
12. Men: Men who agree to abstain from heterosexual intercourse or use contraception and also agree not to donate sperm, as defined below:

    1. If the female partner is of childbearing potential, male patients must abstain from heterosexual intercourse during the treatment period and for 6 months after the last dose of the study drug or use a condom plus another contraceptive method to achieve a contraceptive failure rate of <1% per year. During the same period, male patients must also agree not to donate sperm. If the female partner is already pregnant, male patients must abstain from heterosexual intercourse or use a condom for contraception during the treatment period and for 6 months after the last dose of the study drug to avoid potential effects on the fetus.
    2. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial, patients' preferred lifestyle, and daily activities. Periodic abstinence methods (such as calendar-based methods, ovulation period methods, symptothermal methods, or post-ovulation methods) and withdrawal are not acceptable contraceptive methods.

Exclusion Criteria:

According to the information provided, the following patients are not eligible for participation in this study.

1. Patients with a previous histological/cytological diagnosis of fibrolamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma, or other similar components.
2. Patients with a history of malignancies other than hepatocellular carcinoma, unless they meet the following criteria:

   1. Patients who have undergone potentially curative treatment and have no evidence of the disease within the past 5 years.
   2. Patients who have successfully undergone resection of basal cell carcinoma, squamous cell carcinoma, superficial bladder cancer, cervical carcinoma in situ, or other in situ carcinomas; or patients who have been treated for superficial bladder cancer, have undergone surgical treatment, and have prostate-specific antigen (PSA) tumor markers within the normal range.
3. Patients who are concurrently taking medications that may prolong the QTc interval and/or induce torsades de pointes (Tdp) or medications that affect drug metabolism.

   Patients with a known or suspected history of allergies to sorafenib, lenvatinib, donafenib, or similar drugs.
4. Patients with active bleeding or coagulation abnormalities, bleeding tendencies, or those undergoing thrombolysis, anticoagulant therapy, or antiplatelet therapy.
5. Patients who have experienced thrombosis or thromboembolic events within the past 6 months, such as stroke and/or transient ischemic attack, deep vein thrombosis, pulmonary embolism, etc.

7.Patients who have experienced esophageal or gastric variceal bleeding due to portal hypertension within the past 6 months or any life-threatening bleeding event within the past 3 months. Patients with a history of gastrointestinal bleeding within the past 6 months or clear evidence of gastrointestinal bleeding tendencies, such as high-risk esophageal varices, locally active gastrointestinal ulcers, fecal occult blood ≥(++), are not eligible for inclusion. If fecal occult blood is (+), a gastroscopy examination is required. Evidence or history of bleeding mechanism disorders with ≥3 grade (CTC-AE 5.0) bleeding events, etc.

8.Patients with clinically significant cardiovascular diseases, including but not limited to acute myocardial infarction within the past 6 months, severe/unstable angina or coronary artery bypass grafting, congestive heart failure (NYHA class >2), poorly controlled or requiring pacemaker therapy for arrhythmias, poorly controlled hypertension (systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg) despite medication.

9.Other significant clinical and laboratory abnormalities that the investigator deems to impact safety assessment, such as uncontrolled diabetes, chronic kidney disease, peripheral neuropathy of grade II or higher (CTCAE V5.0), thyroid dysfunction, etc.

10.Active or poorly controlled severe infections, including:

1. HIV-positive (HIV1/2 antibody).
2. Active hepatitis B (positive for HBsAg or HBV DNA>2000 IU/ml and abnormal liver function).
3. Active hepatitis C (positive for HCV antibody or HCV RNA≥103 copies/ml and abnormal liver function).
4. Active tuberculosis.
5. Other uncontrolled active infections (CTCAE V5.0 >2 grade). 11.Patients who have not yet recovered from surgery, with unhealed wounds or severe postoperative complications.

   12.Patients with substance abuse or any medical, psychological, or social conditions that may affect the study, patient compliance, or potentially endanger patient safety.

   13.Patients who have received treatment with potent CYP3A4 inhibitors (such as clarithromycin, indinavir, ketoconazole, lopinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telaprevir, voriconazole, etc.) within 7 days prior to study participation or potent CYP3A4 inducers (such as phenytoin, phenobarbital, primidone, carbamazepine, rifampin, rifabutin, rifapentine, St. John's wort, etc.) within 12 days prior to study participation.

   14.Recipients of multiorgan transplantation. 15.Development of distant metastasis within 1 month after transplantation. 16.Participation in another clinical trial within the past 30 days. 17.Incomplete treatment duration of less than 3 months. 18.The investigator's comprehensive judgment deems the patient unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
EFFICACY: One-year recurrence-free survival rate (1-year RFS rate) | Baseline up to 12 months
  One-year recurrence-free survival rate (1-year RFS rate): The one-year recurrence-free survival rate represents the proportion of patients, within a specified study population, who remain free from disease recurrence for at least one year following a designated treatment or intervention.

SECONDARY OUTCOMES:
EFFICACY: Recurrence-free survival (RFS) duration | Baseline up to approximately 12 months
  Recurrence-free survival (RFS) duration: From randomization to the time of disease recurrence evidence or any cause-induced mortality.
EFFICACY: Overall survival (OS) | Baseline up to approximately 3 years
  Overall survival (OS): The duration from randomization to mortality caused by any underlying factors serves as a crucial metric for evaluating the impact of interventions on study participants.
EFFICACY: Two-year and three-year RFS rates | Baseline up to approximately 2-3 years
  Two-year and three-year RFS rates: The two-year and three-year RFS rate represents the proportion of patients, within a specified study population, who remain free from disease recurrence for at least two or three year following a designated treatment or intervention.
EFFICACY and SAFETY: Graft survival | Baseline up to approximately 3 years
  Graft survival: The interval between the commencement of randomization and the occurrence of graft loss is a pivotal time frame in transplantation research. In cases where patients are unaware of graft loss or when graft loss is not documented upon patient demise without confirmed graft loss, the time of graft loss is retrospectively evaluated using either the date of the last documented contact or the date of death.
QUALITY OF LIFE：Quality of life evaluation | Baseline up to approximately 3 years
  Quality of life evaluation (QoL) according by FACT-Hep.
SAFETY: Incidence of adverse events and serious adverse events | Baseline up to approximately 3 years
  Incidence of adverse events and serious adverse events. Grade by CTCAE 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: haitao zhao, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Chinese Academy of Medical Sciences & Peking Union Medical College Hospital (CAMS&PUMCH), Beijing, Beijing Municipality, China